CLINICAL TRIAL: NCT05040100
Title: Utilizing a 3D Printed Model of the Mediastinum to Teach Thoracic Anatomy to Medical Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natalie Lui, ASSISTANT PROFESSOR OF CARDIOTHORACIC SURGERY, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 52539
Record Dates: First submitted 2021-08-18; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Anatomy Teaching Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded grader scored all tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Textbook Cohort (No Intervention): Trainees underwent a 10-minute lecture using two-dimensional (2D) images of the mediastinum selected from standard textbook resources. The lecture carefully reviewed the mediastinal anatomy reflected in the prosected cadaver and provided a variety of 2D axial, coronal, and sagittal images.
- 3D Model Cohort (Experimental): Trainees underwent a 10-minute lecture using two-dimensional (2D) images of the mediastinum selected from standard textbook resources. The lecture carefully reviewed the mediastinal anatomy reflected in the prosected cadaver and provided a variety of 2D axial, coronal, and sagittal images. Upon completion of the didactic session, the 3D model cohort was provided with an additional 10-minute interactive lecture reviewing the same focused mediastinal anatomical structures using the 3D model.
  Interventions: Other: 3D Mediastinum Model

INTERVENTIONS:
Other: 3D Mediastinum Model — The 3D model cohort was provided with an additional 10-minute interactive lecture reviewing the same focused mediastinal anatomical structures using the 3D model.
  Arms: 3D Model Cohort

SUMMARY:
Three-dimensional (3D) printed anatomic models are increasingly being developed for medical education. The investigators sought to compare the efficacy of a 3D printed model of the mediastinum as a study tool with standard textbooks for teaching medical trainees thoracic anatomy.

Participants were randomly assigned to either a lecture using a standard anatomy textbook or the same lecture along with a 3D printed model of the mediastinum. Participants took a timed pre-test and post-test, identifying 12 mediastinal structures on a prosected human cadaver. Independent and dependent t-tests were used to compare individual and group improvements respectively. A subjective assessment was also performed.

ELIGIBILITY:
Inclusion Criteria:

* Medical trainee

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement from pre-test to post-test | Up to 1 year
  Participants took a same-day timed pre-test and post-test, identifying 12 mediastinal structures on a prosected human cadaver. Independent and dependent t-tests were used to compare individual and group improvements respectively

SECONDARY OUTCOMES:
Subjective Evaluation | Up to 1 year
  Medical trainees were given a subjective assessment on the perceived benefit of the model

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Lui, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States